CLINICAL TRIAL: NCT00031590
Title: Study Of Reduced Dose Craniospinal Radiotherapy (1800 cGy) And Chemotherapy In Children With Newly-Diagnosed Standard-Risk Posterior Fossa Primitive Neuro-ectodermal Tumor (PNET/Medulloblastoma)
Brief Title: Low-Dose Radiation and Combination Chemotherapy Following Surgery in Children With Newly Diagnosed Medulloblastoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated prematurely due to slow accrual.
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Stanford University (Other); Emory University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00-002301; CHP-693 (Other: Children's Hospital of Philadelphia)
Record Dates: First submitted 2002-03-08; First posted 2003-01-27 (Estimated); Results first posted 2019-04-25 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Brain Tumors; Central Nervous System Tumors; Medulloblastoma
Keywords: average risk medulloblastoma; craniospinal radiotherapy; newly diagnosed
MeSH Terms: conditions — Brain Neoplasms; Central Nervous System Neoplasms; Medulloblastoma | interventions — Cisplatin; Platinum; Cyclophosphamide; Etoposide; Lomustine; Vincristine; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study Treatment (Experimental): All subjects will undergo routine surgical staging of their tumor. Treatment must begin within 28 days of surgery. Craniospinal Radiation therapy will last for 6 weeks, five days per week. Once a week during radiation, subjects will also be treated with vincristine. 4 weeks after radiation and vincristine treatment is completed, all subjects will begin 9 cycles (each cycle lasts 6 weeks) of "maintenance chemotherapy" which will be given as 2 different drug combinations, Regimen A (Lomustine, Vincristine, and Cisplatin) and Regimen B (Cyclophosphamide, given with Mesna, and Etoposide [IV and oral]) which will be given in the following order: AABAABAAB (total of 54 weeks).
  Interventions: Drug: Cisplatin; Drug: Cyclophosphamide; Drug: Etoposide; Drug: Lomustine; Drug: Vincristine; Radiation: Craniospinal Radiation

INTERVENTIONS:
Drug: Cisplatin — Given at a dose of 70mg/m2 by intravenous (IV) infusion over 8 hours on day 0 of each cycle (Regimen A only).
  Other Names: CDDP; Platinum
Drug: Cyclophosphamide — Given at a dose of 1g/m2/day by IV infusion on days 0 and 1 of a 6-week cycle. Administration of cyclophosphamide will always be preceded by prehydration and Mesna (Regimen B only).
  Other Names: Cytoxan
Drug: Etoposide — Given at a dose of 150mg/m2/day by IV infusion on days 0 and 1 of a 6-week cycle. Given orally at a dose of 50mg/m2 as a single daily dose for 21 days beginning on day 14 of a cycle (Regimen B only).
  Other Names: VP-16
Drug: Lomustine — Given at a dose of 75mg/m2 taken orally on days 0 of each 6-week cycle with vincristine and cisplatin (Regimen A only).
  Other Names: CCNU
Drug: Vincristine — Given at a dose of 1.5mg/m2 given by IV infusion once a week for the first six weeks of treatment during radiation therapy. During maintenance therapy, it will be given as an IV push on days 0, 7 and 14 of each 6-week cycle (Regimen A only).
  Other Names: Oncovin
Radiation: Craniospinal Radiation — Craniospinal radiation will begin within 28 days of surgery. Craniospinal Radiation therapy will last for 6 weeks, five days per week. Once a week during radiation, subjects will also be treated with chemotherapy (vincristine).
  Other Names: Radiation

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells, but also damages normal cells in the developing brains of children. Combining low-dose radiation therapy in combination with chemotherapy should be effective in treating medulloblastoma while avoiding the long-term side effects of giving higher dose radiation to children with newly diagnosed average risk medulloblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* By giving reduced dose craniospinal radiation followed by nine cycles of maintenance chemotherapy comprised of alternating cycles of lomustine, cisplatin, and vincristine alternating with cyclophosphamide and etoposide, we will reduce the late effects of higher dose radiation in children while maintaining the therapeutic efficacy (86% 3-year relapse-free survival) of current standard therapy
* To evaluate the late neurotoxic effects of low-dose craniospinal radiotherapy, in terms of cognitive, endocrinologic, and auditory function, in these patients.

OUTLINE: This is a multi center study of reduced dose craniospinal radiotherapy and chemotherapy in patients ages 3 - 30 years with newly diagnosed average risk medulloblastoma.

* Induction chemoradiotherapy: Beginning within 28 days after complete surgical resection, patients undergo radiotherapy to the craniospinal axis (1800 centigray (cGy)) followed by conformal radiotherapy to the tumor bed (5400 cGy). Patients receive vincristine weekly for 6 weeks.
* Maintenance chemotherapy: Beginning 4 weeks after the completion of craniospinal radiation therapy, patients receive two 6-week courses of regimen A as outlined below alternating with one 6-week course of regimen B for a total of 9 courses (AABAABAAB).

  * Regimen A: Patients receive oral lomustine and cisplatin on day 0 and vincristine on days 0, 7, and 14.
  * Regimen B: Patients receive cyclophosphamide on days 0 and 1 and etoposide intravenous (IV) on days 0 and 1, followed by oral etoposide on days 14-34.

Patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter with surveillance neuroimaging using Magnetic Resonance Imaging Scan (MRI scan) and clinical examination.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study within 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed medulloblastoma
2. Standard-risk disease
3. No residual tumor greater than 1.5 cm^2 after resection by postoperative MRI

   * No tumor in the spinal or cerebral subarachnoid space by MRI
   * No tumor in the subarachnoid space by Cerebrospinal fluid (CSF)
   * No failure to perform staging studies (spine MRI and CSF cytology) preoperatively or postoperatively
4. Must begin radiotherapy on study within 28 days after surgery

Exclusion Criteria:

1. Prior radiotherapy and anti-tumor chemotherapy other than corticosteroids are not allowed.
2. Pregnant females will not be eligible
3. Patients must begin radiotherapy on protocol within 28 days of completion of surgery. Exceptions need to be approved by the Principal Investigator.
4. Patients with the following will not be eligible:

   * > 1.5cm3 residual tumor following resection as indicated by post-operative MRI.
   * tumor in spinal or cerebral subarachnoid space either by MRI of brain and spine
   * tumor in subarachnoid space by CSF cytology
   * failure to perform staging studies (spine MRI, CSF cytology) either pre- or post- operatively

Ages: 3 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2001-04; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter C. Phillips, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (3):
- United States (3):
  - Lucile Packard Children's Hospital at Stanford University Medical Center, Palo Alto, California
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Minturn JE, Mochizuki AY, Partap S, Belasco JB, Lange BJ, Li Y, Phillips PC, Gibbs IC, Fisher PG, Fisher MJ, Janss AJ. A Pilot Study of Low-Dose Craniospinal Irradiation in Patients With Newly Diagnosed Average-Risk Medulloblastoma. Front Oncol. 2021 Sep 2;11:744739. doi: 10.3389/fonc.2021.744739. eCollection 2021. PMID 34540703

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at three participating institutions namely Childrens Hospital of Philadelphia, Stanford University and Emory University.
Pre-assignment Details: Thirty subjects signed consent. One subject was deemed ineligible due to positive cerebrospinal fluid (CSF) and second subject was declared ineligible due to delayed start of radiation therapy (RT). Remaining 28 subjects continued on study.
Groups:
- Study Treatment: All subjects will undergo routine surgical staging of their tumor. Treatment must begin within 28 days of surgery. Craniospinal Radiation therapy will last for 6 weeks, five days per week. Once a week during radiation, subjects will also be treated with vincristine. 4 weeks after radiation and vincristine treatment is completed, all subjects will begin 9 cycles (each cycle lasts 6 weeks) of "maintenance chemotherapy" which will be given as 2 different drug combinations, Regimen A (Lomustine, Vincristine, and Cisplatin) and Regimen B (Cyclophosphamide, given with Mesna, and Etoposide) which will be given in the following order (total of 54 weeks):1st-Regimen A, 2nd-Regimen A, 3rd-Regimen B, 4th-Regimen A, 5th-Regimen A, 6th-Regimen B, 7th-Regimen A, 8th-Regimen A, 9th-Regimen B. Cisplatin: Given at a dose of 70mg/m2 by intravenous (IV) infusion over 8 hours on day 0 of each cycle (Regimen A only). Cyclophosphamide: Given at a dose of 1g/m2/day by IV infusion on days 0 and 1 of a 6
Period: Overall Study
Arm/Group | Study Treatment
Started | 28
Completed | 25
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Withdrawal by parents | 2

BASELINE CHARACTERISTICS:
Arm/Group | Study Treatment
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 28
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 19
Race/Ethnicity, Customized [Number; unit: participants]
  White | 17
  African american | 5
  Asian | 1
  Hispanic | 5
  Other | 0
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Evaluate Rate of Late Neurotoxic Effects
Description: Evaluate the late neurotoxic effects of low dose craniospinal radiation, including neurocognitive decline as measured by serial neurocognitive testing.
Time Frame: 3 years
Population: The primary endpoint was not met due to lack of evaluable data from non-compliance with neurocognitive testing. Baseline neurocognitive testing was performed on 5 of 28 (18%) of study subjects. Of those 5 subjects with baseline testing, only 1 completed follow up neurocognitive testing at the protocol specified time points.
Groups:
- Study Treatment: All subjects will undergo surgical resection and routine staging (MRI spine and LP for CSF cytology). Subjects aged 3-30 yrs with M0 disease are eligible. Treatment must begin within 28 days of surgery. Reduced dose craniospinal irradiation (CSI) (1800 centiGray (cGy) CSI + 3780 cGy tumor bed) will last for 6 weeks with concurrent, weekly vincristine. 4 weeks after radiation therapy is completed, all subjects will begin 9 cycles of maintenance chemotherapy: Regimen A (CCNU, Vincristine, and Cisplatin) and Regimen B (Cyclophosphamide, given with Mesna, and Etoposide). Cycles will be given as AABAABAAB
  Regimen A:
  Cisplatin: 70mg/m2/dose x 1 dose on day 0 Vincristine: 1.5 mg/m2/dose on days 0, 7, 14 CCNU: 75 mg/m2/dose x 1 dose on day 0
  Regimen B:
  Cyclophosphamide: 1g/m2/dose on days 0 and 1 Etoposide: 150 mg/m2/dose (IV) on days 0 and 1 Etoposide: 50 mg/m2/day PO on days 14-34 (21 days total)
Arm/Group | Study Treatment
Number analyzed (Participants) | 0

2. Secondary Outcome: Long Term Survival
Description: Survival Endpoints:
  Event free survival and overall survival were assessed at 5 years from time of study enrollment
Time Frame: Up to 5 years from date of randomization until the date of first documented progression or date of death from any cause, whichever came first.
Population: All subjects who received radiation and started chemotherapy.
Measure: Number; unit: Percentage of participants
Groups:
- Study Treatment: All subjects will undergo surgical resection and routine staging (Magnetic Resonance Imagine (MRI) spine and Lumbar Puncture (LP) for cerebrospinal fluid (CSF) cytology). Subjects aged 3-30 yrs with M0 disease are eligible. Treatment must begin within 28 days of surgery. Reduced dose craniospinal RT (1800 cGy CSI + 3780 cGy tumor bed) will last for 6 weeks with concurrent, weekly vincristine. 4 weeks after radiation therapy is completed, all subjects will begin 9 cycles of maintenance chemotherapy: Regimen A (Lomustine (CCNU), Vincristine, and Cisplatin) and Regimen B (Cyclophosphamide, given with Mesna, and Etoposide). Cycles will be given as AABAABAAB
  Regimen A:
  Cisplatin: 70mg/m2/dose x 1 dose on day 0 Vincristine: 1.5 mg/m2/dose on days 0, 7, 14 CCNU: 75 mg/m2/dose x 1 dose on day 0
  Regimen B:
  Cyclophosphamide: 1g/m2/dose on days 0 and 1 Etoposide: 150 mg/m2/dose intravenous (IV) on days 0 and 1 Etoposide: 50 mg/m2/day oral (PO) on days 14-34 (21 days total)
Arm/Group | Study Treatment
Number analyzed (Participants) | 28
Percentage of participants
  5 year Overall Survival (OS) | 87.5
  5 year Event Free Survival (EFS) | 70

ADVERSE EVENTS:
Description: Adverse events were recorded in the following categories: auditory toxicity, renal toxicity, and endocrinologic toxicity
Groups:
- Study Treatment: All subjects will undergo routine surgical staging of their tumor. Treatment must begin within 28 days of surgery. Craniospinal Radiation therapy will last for 6 weeks, five days per week. Once a week during radiation, subjects will also be treated with vincristine. 4 weeks after radiation and vincristine treatment is completed, all subjects will begin 9 cycles (each cycle lasts 6 weeks) of "maintenance chemotherapy" which will be given as 2 different drug combinations, Regimen A (Lomustine, Vincristine, and Cisplatin) and Regimen B (Cyclophosphamide, given with Mesna, and Etoposide) which will be given in the following order (total of 54 weeks):1st-Regimen A, 2nd-Regimen A, 3rd-Regimen B, 4th-Regimen A, 5th-Regimen A, 6th-Regimen B, 7th-Regimen A, 8th-Regimen A, 9th-Regimen B Cisplatin: Given at a dose of 70mg/m2 by intravenous (IV) infusion over 8 hours on day 0 of each cycle (Regimen A only). Cyclophosphamide: Given at a dose of 1g/m2/day by IV infusion on days 0 and 1 of a 6
Arm/Group | Study Treatment
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 28/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Study Treatment (N=28)
hearing loss (Ear and labyrinth disorders) | 15
creatinine clearance (Renal and urinary disorders) | 5
thyroid dysfunction (Endocrine disorders) | 11
growth hormone deficiency (Endocrine disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes